CLINICAL TRIAL: NCT00115713
Title: Comparison of Aerobic Versus Resistance Exercise Training in Enhancing Quality of Life in Early Stage Breast Cancer Survivors Receiving Chemotherapy: A Multi-Centre Randomized Trial
Brief Title: Effects of Aerobic Exercise Versus Weight Training in Breast Cancer Survivors During Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Canadian Breast Cancer Research Alliance (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ETH-02-70-85
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Breast Neoplasms
Keywords: Aerobic Exercise; Weight Lifting; Breast Cancer; Quality of Life
MeSH Terms: conditions — Breast Neoplasms | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Aerobic Exercise Training
Behavioral: Resistance Exercise Training

SUMMARY:
The purpose of this study is to compare the effects of two different types of exercise, aerobic exercise training (AET) and resistance exercise training (RET), on quality of life (QoL) in early stage breast cancer survivors receiving chemotherapy. It is hypothesized that both AET and RET would have beneficial effects on QoL.

DETAILED DESCRIPTION:
The study was a prospective, three-armed, randomized controlled trial. Participants were stratified by site (Edmonton, Ottawa, and Vancouver) and planned chemotherapy protocol (taxane-based versus nontaxane-based) and randomly assigned to AET, RET, or usual care (UC) in a 1:1:1 ratio using a random-numbers table. Participants assigned to the AET group were asked to perform aerobic exercise three times per week on a recumbent or upright cycle ergometer, treadmill, or elliptical. Exercise duration began at 15 minutes for weeks 0 through 2, and then systematically increased by 5 minutes every three weeks thereafter to 45 minutes for weeks 18 and beyond. Exercise intensity began at 60% of VO2max for weeks 0 through 2 and then systematically increased by 10% every 6 weeks thereafter to 80% of VO2max for weeks 12 and beyond. Warm-up and cool-down periods consisted of 5 minutes of aerobic activity at the power output of the ventilatory equivalent for oxygen (approximately 50% of peak oxygen consumption). Participants assigned to the RET group were asked to perform resistance exercise three times per week, which consisted of two sets of 10 repetitions of 9 different exercises performed at 60-70% of 1-repetition maximum. The specific exercises were: leg extension, leg curl, calf raises, chest press, latissimus pulldown, overhead press, triceps extension, biceps curls, and modified curl-ups. Resistance was increased by approximately 10% or the next weight level when the participant was able to complete 12 repetitions per set without difficulty.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer early stage I -IIIA
* Completed axillary surgery
* Scheduled to receive adjuvant chemotherapy for 9 - 24 weeks
* Approval of the treating oncologist
* Able to understand and provide written informed consent in English or French (Ottawa)
* 18+ years of age
* No uncontrolled hypertension, cardiac illness, psychiatric condition
* No contraindication to exercise as determined by a fitness test

Exclusion Criteria:

* Pregnant.
* Unwilling to accept randomization.
* Any medical condition that would be a contraindication to exercise. The clinicians will make this decision.
* Unwilling to travel to/participate in the exercise program as defined by the protocol.
* Previous chemotherapy (previous cancer is NOT an exclusion criteria).
* Cancer recurrence.
* Planned/known absence of greater than 2 weeks during the intended study period.
* Previous therapy for known breast cancer.
* Those who have had TRAM (i.e., Transabdominal Rectus Abdominus Muscle Reconstructive Surgery) done.
* Moderate lymphedema (>20% or >200mL difference between the affected arm and the unaffected arm).

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240
Dates: Start 2003-04; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Quality of Life

SECONDARY OUTCOMES:
Physical Fitness
Body Composition
Lymphedema
Treatment Completion Rates
Selected Biomarkers
Exercise Adherence Rates and Determinants

CONTACTS AND LOCATIONS:
Overall Officials: Kerry S Courneya, PhD, Principal Investigator — University of Alberta
Locations (3):
- Canada (3):
  - University of Alberta, Edmonton, Alberta
  - University of British Columbia, Vancouver, British Columbia
  - Ottawa Hospital, Ottawa, Ontario

REFERENCES:
- [Derived] An KY, Arthuso FZ, Kang DW, Morielli AR, Ntoukas SM, Friedenreich CM, McKenzie DC, Gelmon K, Mackey JR, Courneya KS. Exercise and health-related fitness predictors of chemotherapy completion in breast cancer patients: pooled analysis of two multicenter trials. Breast Cancer Res Treat. 2021 Jul;188(2):399-407. doi: 10.1007/s10549-021-06205-8. Epub 2021 Mar 29. PMID 33779887
- [Derived] Courneya KS, Segal RJ, McKenzie DC, Dong H, Gelmon K, Friedenreich CM, Yasui Y, Reid RD, Crawford JJ, Mackey JR. Effects of exercise during adjuvant chemotherapy on breast cancer outcomes. Med Sci Sports Exerc. 2014 Sep;46(9):1744-51. doi: 10.1249/MSS.0000000000000297. PMID 24633595
- [Derived] Dolan LB, Gelmon K, Courneya KS, Mackey JR, Segal RJ, Lane K, Reid RD, McKenzie DC. Hemoglobin and aerobic fitness changes with supervised exercise training in breast cancer patients receiving chemotherapy. Cancer Epidemiol Biomarkers Prev. 2010 Nov;19(11):2826-32. doi: 10.1158/1055-9965.EPI-10-0521. Epub 2010 Sep 22. PMID 20861399
- [Derived] Courneya KS, Reid RD, Friedenreich CM, Gelmon K, Proulx C, Vallance JK, McKenzie DC, Segal RJ. Understanding breast cancer patients' preference for two types of exercise training during chemotherapy in an unblinded randomized controlled trial. Int J Behav Nutr Phys Act. 2008 Oct 27;5:52. doi: 10.1186/1479-5868-5-52. PMID 18954442